CLINICAL TRIAL: NCT06125652
Title: Application of Anti Tim-3/CD123 CAR-T Cell Therapy in Relapsed and Refractory Acute Myeloid Leukemia (rr/AML)
Brief Title: Administration of Anti Tim-3/CD123 CAR-T Cell Therapy in Relapsed and Refractory Acute Myeloid Leukemia (rr/AML)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, President, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2023-KL358-01
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti Tim-3/CD123 CAR-T cell therapy (Experimental): Enrolled patients will receive prespecified dose of autologous CAR-T cells.
  Interventions: Drug: anti Tim-3/CD123 CAR-T cell therapy

INTERVENTIONS:
Drug: anti Tim-3/CD123 CAR-T cell therapy — Enrolled patients will receive prespecified dose of autologous CAR-T cells.

SUMMARY:
To evaluate the safety and efficacy of anti Tim3/CD123 CAR-T cells in the treatment of relapsed and refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Cluster of Differentiation 123 (CD123) is usually overexpressed on leukemia stem cells (LSCs) in acute myeloid leukemia (AML). However, CD123 has poor specificity and is also expressed on normal hematopoietic stem cells (HSC), myeloid cells, and some non-hematopoietic cells. This leads to widespread on-target off-tumor effect in the clinical application of anti CD123 CAR-T cells, manifested as severe bone marrow suppression, organ damage, and patients experiencing infections, bleeding, and organ dysfunction. T cell immunoglobulin and mucin domain 3 (Tim-3) belongs to the Tim gene family. 85% of LSCs highly express Tim-3, while normal hematopoietic stem/progenitor cells (HSC/P), granulocytes, and macrophages do not express Tim-3. Compared with CD123, seeing Tim-3 as a recognition tool for LSCs has higher specificity. In vivo and in vitro studies have confirmed that anti Tim-3 CAR-T cells have significant anti LSCs effects, while not affecting the ability of normal HSC/P to form colonies and differentiate lineages. We believe that using both Tim-3 and CD123 as targets for CAR-T cells can improve the specificity of recognizing LSCs, reduce the killing effect of CAR-T cells on HSC/P expressing CD123, and thus reduce the on-target off-tumor effect.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must sign and date the Informed Consent before initiating any study specific procedures or activities;
2. At the age of 18-70 years old;
3. Diagnosed as relapse/refractory (r/r) de novo or secondary acute myeloid leukemia (AML);
4. The patient has recovered from the toxicity of previous treatment;
5. ECOG score ≤ 2 and expected survival period is not less than 3 months;
6. Adequate organ function defined as:AST ≤3×ULN; ALT ≤3×ULN; Total bilirubin ≤1.5×ULN; Serum creatinine ≤1.5×ULN, or CCR≥60 mL/min; Hemoglobin ≥60g/L ; Indoor oxygen saturation ≥92%; LVEF≥45%;
7. Pregnancy testing: females of childbearing potential must have a negative serum or urine pregnancy test;
8. From the use of study drug to 2 years after treatment, males and female of childbearing potential must agree to use an effective method of contraception.

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia;
2. History or presence of a CNS disorder;
3. HBsAg is positive; HCV #HIV or Syphilis antibody are positive, CMV-DNA in peripheral blood is more than≥500 copies /mL;
4. History of severe hypersensitivity reaction;
5. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, atrial fibrillation, or other clinically significant cardiac disease within 12 months before enrollment;
6. History of organ transplant surgery;
7. Required systemic application of immunosuppressive or other drugs;
8. Auto-SCT within the 3 months before enrollment;
9. Active autoimmune or inflammatory diseases of the nervous system (e.g., Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES));
10. Requirement for urgent therapy due to ongoing or impending oncologic emergency (eg, leukostasis or tumor lysis syndrome (TLS)) ;
11. Presence or suspicion of a fungal, bacterial, viral, or other infection that is uncontrolled or requiring antimicrobials for management;
12. Live vaccine received within the ≤ 4 weeks before enrollment;
13. Persons with serious mental illness;
14. History of major surgical operations four weeks before enrollment;
15. History of alcoholism or substance abuse;
16. Was identified by the investigators as unsuitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity #DLT# | Baseline up to 28 days after CAR-T cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
MRD negative overall response rate (MRD- ORR) | 3 months
  Assessment of MRD negative overall response rate (MRD- ORR) at 3 months of treatment
Overall response rate (ORR) | Month 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi ) at Month 6, 12, 18 and 24
Event-free survival (EFS) | Month 6, 12, 18 and 24
  Assessment of EFS at Month 6, 12, 18 and 24
Overall survival (OS) | Month 6, 12, 18 and 24
  Assessment of OS at Month 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, MD.,PD., Study Chair — The Affiliated Hospital oh Xuzhou Medical University
Locations (1):
- Kailin Xu, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No